CLINICAL TRIAL: NCT05946239
Title: Evaluating the Manage My Pain App in Pain Clinics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Ontario Bioscience Innovation Organization (Unknown); Alberta Health services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro00126058
Record Dates: First submitted 2023-07-07; First posted 2023-07-14 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Pain
Keywords: pain management; digital health; communication; quality of life; chronic pain; psychology; chronic disease management; anxiety; medication usage; patient oriented research
MeSH Terms: conditions — Pain; Agnosia; Communication; Chronic Pain; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: A randomized controlled trial (RCT) using quantitative approaches will be undertaken to assess the impact of MMP on chronic pain clinic waitlist patient health outcomes prior to attending their first pain clinic appointment. This study will have 1 intervention group (access to MMP + standard care) and 1 control group (standard care). Participants will be randomly assigned to the intervention group or control group at a 2:1 ratio to account for variations in App usage.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manage My Pain App Intervention (Experimental): Participants will have access to the MMP App and standard care for 60 days.
  Interventions: Other: Manage My Pain App
- Control Group (No Intervention): Participants will engage in standard care for 60 days.

INTERVENTIONS:
Other: Manage My Pain App — This digital application helps patients measure, track, and manage chronic pain, functionality, and medication use. MMP can also be used to share patient pain experiences with their circle of care via reports and offers educational resources for patients.
  Arms: Manage My Pain App Intervention

SUMMARY:
Chronic Pain is one of the most common reasons adults seek medical care, and has been linked to restrictions in mobility and daily activities, dependence on opioids, anxiety and depression, and poor perceived health or reduced quality of life. Chronic Pain Clinics are an effective solution, however, the resources available and investments have fallen behind the growing needs of patients. Local waitlists have thousands of patients with wait times between 1 to 3 years, with many receiving little to no specialized support while waiting. Tools and technology that can help patients and healthcare providers understand and manage the patients' pain are needed for the effectiveness of the healthcare system.

In response to this problem, the Manage My Pain (MMP) App, which allows patients to log daily reflections of functionality, pain, and medication use; as well as, provide educational resources is a potential support for patients on the waitlist. This log is intended to support the patient understanding and management of their pain, and share their reports with their circle of care.

This study will assess the impact of MMP on waitlist patients' health outcomes compared to a control group of waitlist patients over 60 days.

DETAILED DESCRIPTION:
Chronic Pain is one of the most common reasons adults seek medical care and has been linked to restrictions in mobility and daily activities, dependence on opioids, anxiety, depression, and poor perceived health or reduced quality of life. Currently, local pain clinic waitlists have thousands of patients with wait times between 1 to 3 years, with many receiving little to no specialized support while waiting for an appointment. To address this problem, this study assesses the impact of the MMP App to support the health and medication use of patients on the waitlist. Using this approach patients on the waitlist can use this app to report their pain, functionality, reflections, and medication use, as well as read educational resources about pain management.

This study tests the effectiveness of the MMP App versus a control group (i.e., standard practice) on health outcomes and mediation use over 60 days in a randomized control trial (RCT). The primary outcomes are pain, anxiety, pain self-efficacy, and quality of life. Secondary outcome is medication usage. Researchers will use descriptive and regression analysis to assess the data collected.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* On the Calgary Pain Clinic waitlist

Exclusion Criteria:

* Participants were excluded if they did not meet any of the above criteria
* Patients declining or unable to complete the consent process for the study
* No internet access
* No access to a device or computer to display the app/website

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2023-07-10 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
EuroQol-5 Dimension-5 Levels (EQ5D5L) | 60 days
  EQ5D5L is a short descriptive questionnaire and a visual analogue scale that are simple to complete and assess five dimensions of quality of life including: mobility, selfcare, usual activities, pain/discomfort, and anxiety and depression (EuroQol, 2019). Each quality of life dimension will be assessed according to the following five level response scale, which varies in degree of severity from: no problem, light problem, moderate problems, severe problems, and unable to / extreme problems (EuroQol, 2019). The respondent will be asked to select the response item that most appropriately matches their current state (EuroQol, 2019). The single item score for each dimension is used assess the dimension, rather than a composite score. This instrument has been proven to be valid, reliable, and responsive in numerous conditions and populations (EuroQol, 2019; Finch et al., 2018).
Generalized Anxiety Disorder (GAD-7) | 60 days
  The GAD-7 is a brief self-report assessment of anxiety severity for clinical practice and research (Spitzer et al., 2006). The GAD-7 consists of 7-items assessing anxiety on a four-point scale with response options including: not at all (score=0), several days (score=1), more than half the days (score=2), and nearly every day (score=3). To obtain the GAD-7 score, all scores are added to develop a total anxiety score. A score of 0 to 4 = minimal anxiety, 5 to 9 = mild anxiety, 10 to 14 = moderate anxiety, and a score greater than 15 = severe anxiety (Plummer et al., 2016). To screen for anxiety disorders, a score of 8 or greater represents a reasonable cut-point for identifying probable cases of generalized anxiety disorder (Plummer, et al 2016). The GAD-7 has been demonstrated to be a reliable and valid tool to detect generalized anxiety (Spitzer et al., 2006).
Pain (Numeric Pain Rating Scale) | 60 days
  The Pain Numeric Rating Scale (NRS) is an 11 point scale that asks patients to identify the number between 0 (no pain at all) and 10 (the worst pain ever possible) that fits their pain intensity (McCaffery & Beebe, 1989).
Pain self-efficacy (PSEQ-4) | 60 days
  PSEQ-4 is an instrument to assess pain self-efficacy for clinical and research purposes (Chiarotto et al., 2016). The PSEQ-4 includes four items scored on a 7-point Likert scale ranging from not at all confident (score=0) to completely confident (score=6). Pain self-efficacy is calculated by summing the scores to determine a total score ranging from 0 to 24 (Chiarotto et al., 2016). High scores indicate greater pain self-efficacy. A systematic review has found that the PSEQ-4 has demonstrated excellent validity, reliability, and responsiveness among chronic lower back pain patients (Dubé et al., 2021). The PSEQ-4 may replace the full PSEQ and have similar responsiveness (Chiarotto et al., 2016).

SECONDARY OUTCOMES:
Medication Usage | 60 days
  A medication usage questionnaire used in pain clinics was modified with clinicians for this study. The survey asks if any of the listed medication (i.e.,Tramadol, Acetaminophen/ Codeine (Tylenol No 3, Hydromorphone, Hydromorphone Contin, Oxycodone 5mg/ Acetaminophen 325mg (Percocet), Oxycodone 5mg/Naloxone 10mg (Targin), Oxycodone, Oxycontin, Codeine, Morphine, Morphine Contin, Oxycodone, Oxycontin, Methadone, Fentanyl, Buprenorphine, Other Opioid) were taken in the last 7 days. If the medication was taken, the dose and frequency of administration was recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Calgary Chronic Pain Centre, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chiarotto A, Vanti C, Cedraschi C, Ferrari S, de Lima E Sa Resende F, Ostelo RW, Pillastrini P. Responsiveness and Minimal Important Change of the Pain Self-Efficacy Questionnaire and Short Forms in Patients With Chronic Low Back Pain. J Pain. 2016 Jun;17(6):707-18. doi: 10.1016/j.jpain.2016.02.012. Epub 2016 Mar 11. PMID 26975193
- [Background] Dube MO, Langevin P, Roy JS. Measurement properties of the Pain Self-Efficacy Questionnaire in populations with musculoskeletal disorders: a systematic review. Pain Rep. 2021 Dec 21;6(4):e972. doi: 10.1097/PR9.0000000000000972. eCollection 2021 Nov-Dec. PMID 34963996
- [Background] Finch AP, Brazier JE, Mukuria C. What is the evidence for the performance of generic preference-based measures? A systematic overview of reviews. Eur J Health Econ. 2018 May;19(4):557-570. doi: 10.1007/s10198-017-0902-x. Epub 2017 May 30. PMID 28560520
- [Background] Haefeli M, Elfering A. Pain assessment. Eur Spine J. 2006 Jan;15 Suppl 1(Suppl 1):S17-24. doi: 10.1007/s00586-005-1044-x. Epub 2005 Dec 1. PMID 16320034
- [Background] Plummer F, Manea L, Trepel D, McMillan D. Screening for anxiety disorders with the GAD-7 and GAD-2: a systematic review and diagnostic metaanalysis. Gen Hosp Psychiatry. 2016 Mar-Apr;39:24-31. doi: 10.1016/j.genhosppsych.2015.11.005. Epub 2015 Nov 18. PMID 26719105
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Pain: clinical manual for nursing practice Pain: clinical manual for nursing practice Margo McCaffery Alexander Beebe Mosby Yearbook UK pound17.25 0 7234 1992 2. Nurs Stand. 1994 Dec 7;9(11):55. doi: 10.7748/ns.9.11.55.s69. PMID 27527475
- See also: EuroQol Research Foundation. (2019). EQ5D5L User Guide — https://euroqol.org/publications/user-guides/